CLINICAL TRIAL: NCT04174690
Title: Development of Balance Analysis System Through Biaxial Rotation Force Platform Posturography Combined With Electromyography
Brief Title: Balance Analysis System Through Biaxial Rotation Force Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Terigi Augusto Scardovelli, Principal Investigator, University of Mogi das Cruzes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02651118.0.0000.5497
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2019-11

CONDITIONS: Balancing Interference
Keywords: Center of pressure; Dynamic postural balance; Force platform; Posturography; Electromyography

STUDY DESIGN:
Intervention Model Description: Biaxial rotation force platform combined with electromyography
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance (Experimental): Volunteers aged from 18 years to over 60 years were selected without compromise. The tests were performed in a single session lasting 1 hour where the volunteers will do the tests on the force platform.
  Interventions: Device: Force platform

INTERVENTIONS:
Device: Force platform — In order to volunteers to be selected for collection a recruitment test will be taken, the volunteer will have to stand on one foot for 5 seconds without additional support. So that the volunteer can go to the balance test on the force platform, he will be dressed with safety equipment (harness), and will also have the attachment of the electrodes.

SUMMARY:
This study developed a system for studying an individual's postural balance in an upright position on a force platform with controlled movement of 2-axis rotation (transverse and anteroposterior), by analyzing lower limb muscle activation and data from Pressure Center of displacement.

DETAILED DESCRIPTION:
The use of rotating force platforms has proven to be an important resource in the study of postural balance and motor control. Platforms composed of two force plates allow the analysis of the load relationship between the feet and the study of the coordination of the lower body segments in postural control. Center of pressure displacement data during perturbations generated by platform rotation allow the study of dynamic postural balance. However, devices that meet these characteristics are not common and have limitations on amplitude or speed of rotation. Thus, a force platform composed of two plates was developed, capable of collecting data for the calculation of the parameters of the center of pressure, differentiating each foot, with a computerized system to control amplitude and speed of rotation in the mid-lateral and anteroposterior axes. A new version of embedded and supervisory systems that control the device, collect and process the created data has also been developed. For platform functionality tests, volunteers were divided into three groups of 15 individuals: Group 1 (G1): women aged 18 to 40 years; Group 2 (G2): women aged 40 to 60 years; Group 3 (G3): women over 60 years old.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Ages 18 to 80 years
* Asymptomatic
* Resident of the city of mogi das cruzes.
* You will have to sign the consent form

Exclusion Criteria:

* History of dizziness or dizziness crisis not explained in the last year;
* Any musculoskeletal or neurological disorders;
* Significant pain that limits daily functions;
* Known uncorrected vestibular problems.
* Fall History

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Center of pressure offset | 1 hour
  With the volunteer allocated on the platform in an upright position with the malleoli aligned with the central axis of rotation of the platform will be collected the displacement of the center of pressure. Unit of measure: millimeters (mm).

SECONDARY OUTCOMES:
Electromyographic signal | 1 hour
  Electromyographic signal of the anterior tibial and gastrocnemius muscle. unit of measurement in microvolts (µV).

OTHER OUTCOMES:
Speed of movement of center of pressure | 1 hour
  With the volunteer allocated on the platform in an upright position with the malleoli aligned with the central axis of rotation of the platform will be collected the speed of the center of pressure unit of measure: millimeters per second (mm / s).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro P Silva, PhD, Principal Investigator — University of Mogi das Cruzes
Locations (1):
- Alessandro Pereira da Silva, Mogi das Cruzes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No